CLINICAL TRIAL: NCT03236883
Title: Phase I Study of Nonmyeloablative Allogeneic Hematopoietic Stem Cell Transplantation in the Treatment of Pancreatic Cancer
Brief Title: Nonmyeloablative Allogeneic Hematopoietic Stem Cell Transplantation in the Treatment of Pancreatic Cancer
Acronym: HST
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NST-01
Record Dates: First submitted 2017-07-12; First posted 2017-08-02 (Actual); Last update posted 2017-08-02 (Actual); Status verified 2017-04

CONDITIONS: Pancreatic Cancer Stage III; Pancreatic Cancer Stage IV
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- GEM plus GPBSC (Experimental): Gemcitabine chemotherapy with mobilized GPBSC infusion:Gemcitabine 1000mg/m2 +GPBSC(2-3)*10^8/kg
  Interventions: Drug: Gemcitabine; Other: GPBSC
- Gemcitabine (Other)
  Interventions: Drug: Gemcitabine
- GPBSC (Other)
  Interventions: Other: GPBSC

INTERVENTIONS:
Drug: Gemcitabine — Chemotherapy: Gemcitabine is administered Intravenous injection once a week，at a dose of 1000 mg/m2, for 3consecutive weeks,followed by a 7-days rest,repeated every 4weeks,three times in all.
  Arms: GEM plus GPBSC; Gemcitabine
Other: GPBSC — immunotherapy :GPBSC were collected from donor .Cells were infused to the patients in 4 week,at a dose of (2-3)*10^8/kg,once a month,repeated every 4weeks,three times in all.
  Arms: GEM plus GPBSC; GPBSC

SUMMARY:
To evaluate the safety and efficacy of non-myeloablative hematopoietic stem cell transplantation in the treatment of pancreatic cancer.

DETAILED DESCRIPTION:
Allogeneic hematopoietic stem cell transplantation has been successfully used for the treatment of hematopoietic malignancy. In recent years, non-myeloablative hematopoietic stem cell transplantation (NST) has been introduced to treat solid tumors due to the Graft-versus tumor effect. In this study, the investigators try to evaluate the safety and efficacy of NST in the treatment of unresectable pancreatic cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* PET-CT/EUS-FNA cytologically confirmed stage III -Ⅳ of pancreatic cancer
* Between 18 and 80 years old
* Karnofsky Performance Status (KPS) ≥ 70%，Guaranteed treatment for 3 months
* Normal functions of heart, lung and kidney
* Adequate hematological profile： Hemoglobin ≥ 9.0 g/dL、 Absolute granulocyte count ≥ 1,500/mm^3 、Platelet count ≥ 100,000/mm^3， start the treatment within 14 days after these results meet the requirements
* A life expectancy > 3 months
* Informed consent signed
* HLA-haplotype-matched immediate family health donors who have been confirmed by laboratory HLA genotypes
* Interval the last anti-tumor treatment for more than 3 months

Exclusion Criteria:

* Highly allergic or people with severe allergies
* Brain metastasis or Primary central nervous system malignancy
* Suffer from clinical illnesses that affect clinical trials, including but not limited to： Uncontrollable diabetes；active infectious disease or uncontrollable infection; acute and chronic liver disease; confirmation of HIV infection; uncontrollable hypertension, symptomatic congestive heart-failure, unstable angina pectoris, and myocardial infarction, uncontrollable arrhythmia over the last 6 months.
* Combined heart, lung, kidney and other vital organs dysfunction
* A serious coagulation dysfunction, a clear history of other tumors
* Pregnant and lactating women
* Mental illness, affecting the compliance of clinical trials
* The patient will participate in other trials within 10 days prior to the trial or While participating in other tests
* Patients underwent weight loss by 10% and above within 6 weeks before the start of the trial
* Neutrophils<500mm^3 or Platelet count<50,000/mm^3
* Need to drive and manipulate the machine during the trial

Donor's Inclusion Criteria:

* First-degree relatives of patients
* Age<55 years old
* Normal functions of heart, lung and kidney
* Adequate hematological profile： Hemoglobin ≥ 9.0 g/dL、 Absolute granulocyte count ≥ 1,500/mm^3 、Platelet count ≥ 100,000/mm^3、WBC≥ 3000/mm^3， start collecting stem cells within 14 days after these results meet the requirements
* Informed consent signed

Donor's exclusion Criteria:

* Highly allergic or people with severe allergies
* The person who have history of atherosclerosis, venous thrombosis or autoimmune disease
* A serious coagulation dysfunction, a clear history of other tumors
* Infectious disease or carriers
* Pregnant and lactating women
* Mental illness, affecting the compliance of clinical trials
* WBC<4000/mm^3、PLT<70*10^9/L

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-04 (Actual); Primary Completion 2019-04 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
Survival | 3 months
  Survival will be measured at 3 months after transplant.

SECONDARY OUTCOMES:
Progression free survival（PFS） | 3 months
Overall survival (OS) | 3 months
Response rate | 3 months
Adverse Events | 3 months
Karnofsky Performance Status（KPS） | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Jihui Hao, MD, PHD, Principal Investigator — Tianjin Medical University Cancer Institute and Hospital
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality, China